CLINICAL TRIAL: NCT06787391
Title: Reanimation of Shoulder External Rotation in Children with Obestetric Brachial Plexus Palsy Through Neurotization of Spinal Accessory Nerve to Supra- Scapular Nerve
Brief Title: Reanimation of Shoulder External Rotation Via Neurotization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Faraag Abu el wafa Sayed, Assistant Lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neurotization in OBPP
Record Dates: First submitted 2025-01-14; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Nerve Transfer
Keywords: Nerve transfer

STUDY DESIGN:
Intervention Model Description: Measurement of clinical outcome of Reanimation Of Shoulder External Rotation In Children With Obestetric Brachial Plexus Palsy Through Neurotization Of Spinal Accessory Nerve To Supra- Scapular Nerve.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Just one group of patients children with OBPP presented with deficiency of active shoulder External (Active Comparator)
  Interventions: Procedure: Neurotization of Spinal Accessory Nerve To Supra-Scapular in children with OBPP with deficiency of Shoulder External Rotation; Procedure: Neurotization of Spinal Accessory Nerve To Supra-Scapular Nerve

INTERVENTIONS:
Procedure: Neurotization of Spinal Accessory Nerve To Supra-Scapular in children with OBPP with deficiency of Shoulder External Rotation — Neurotization of Spinal Accessory Nerve To Supra-Scapular Nerve in children with OBPP presented with deficiency of Shoulder External Rotation.
Procedure: Neurotization of Spinal Accessory Nerve To Supra-Scapular Nerve — Just to assess clinical outcomes after Neurotization of spinal accessory nerve to Supra-Scapular Nerve in patients with deficiency of Shoulder External Rotation

SUMMARY:
Measurement of clinical outcome after nerve transfer in deficiency of shoulder external rotation in children with OBPP.

DETAILED DESCRIPTION:
Brachial plexus birth injuries (BPBI) occur in 1-2 per 1,000 live births, often resulting from traction on the shoulder during delivery (1). Right-sided injuries are more common due to fetal positioning.(2) BPBI presentations vary, with upper trunk injuries (Erb's palsy) being most frequent, accounting for 45% of cases.(3) These injuries can impair shoulder abduction, external rotation, and arm function ,He can't flex the elbow to partially reache the hand to the mouth (the trumpet sign) .due to suprascapular nerve (SSN) damage, which is prone to stretching due to its fixed attachments.(4)

Erb's palsy affects muscles like the deltoid and biceps, supraspinatus and infraspinatus.(5) . Assessments include testing hand sensation and noting color or trophic changes. Without SSN reconstruction, secondary glenohumeral complications often arise, necessitating surgical interventions like tendon transfers, joint reductions, or osteotomies.(6)

Nerve transfer, such as spinal accessory nerve (SAN) fascicles to the SSN, has shown superior outcomes for restoring shoulder function. The SAN, a pure motor nerve, is well-suited for direct coaptation without interposition grafts.(7).

Surgical approaches include anterior and posterior methods, each with unique benefits. For instance, the anterior approach allows simultaneous brachial plexus exploration and facilitates nerve repair.(8) , while posterior approach prevents double crush phenomenon.(9)

Despite most children recovering spontaneously, 20-30% experience residual deficits (10). Techniques like tension-free SAN-to-SSN repair aim to improve outcomes. This study evaluates the efficacy of SAN transfers in restoring shoulder stability, abduction, and external rotation in BPBI patients.(11)

ELIGIBILITY:
Inclusion Criteria:

* children within 1.5 - 3 years .
* No previous surgery
* full passive ROM
* presented with Trumpet sign

Exclusion Criteria:

* age <1.5 - >3 years
* previous surgery in the shoulder
* Stiff shoulder.
* total OBPP
* traumatic BPI
* follow up <1 year.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Neurotization in OBPP | Baseline
  Improvement in Shoulder External Rotation after neurotization, and Functional Outcome Scores using mallet score Measurement of the clinical outcome of Active shoulder external rotation following Spinal accessory nerve to supra scapular Nerve transfer in children with Obstetric brachial plexus palsy, ,
  * follow up one year or more , or Recovery of active ER .
  * based on:-
    * 1-------- mallet score from 1 to 5:--- (12)
      1. Flail shoulder 2. Zero degree external rotation 3. Active ER up to 20 degrees 4. Active ER over than 20 degrees 5. Normal shoulder
    * 2----Gilbert shoulder score :- for shoulder ROM and strength (13) 0- complete flail shoulder( none)
      1. no active ER , Abduction to 45° ( poor)
      2. neutral ER , Abduction<90(fair)
      3. weak ER , Abduction= 90°( satisfactory)
      4. incomplete ER, Abduction<120°( good )
      5. active ER , Abduction> 120°( excellent)

SECONDARY OUTCOMES:
Measurement of ROM after Neurotization | Baseline
  Asses the recovery of shoulder stability and overall. Shoulder Range of Motion (ROM):

CONTACTS AND LOCATIONS:
Overall Officials: Omar Ahmed Refai Mohammed, Assistant professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elzinga KE, Curran MW, Morhart MJ, Chan KM, Olson JL. Open Anterior Release of the Superior Transverse Scapular Ligament for Decompression of the Suprascapular Nerve During Brachial Plexus Surgery. J Hand Surg Am. 2016 Jul;41(7):e211-5. doi: 10.1016/j.jhsa.2016.03.005. Epub 2016 Apr 22. PMID 27113908
- [Background] Pondaag W, Malessy MJ, van Dijk JG, Thomeer RT. Natural history of obstetric brachial plexus palsy: a systematic review. Dev Med Child Neurol. 2004 Feb;46(2):138-44. doi: 10.1017/s0012162204000258. No abstract available. PMID 14974639
- [Background] Gilbert A. Indications and strategy. In: Gilbert A, editor. Brachial plexus injuries. London: Martin Dunitz; 2001. p. 205-10.
- [Background] Dailiana ZH, Mehdian H, Gilbert A. Surgical anatomy of spinal accessory nerve: is trapezius functional deficit inevitable after division of the nerve? J Hand Surg Br. 2001 Apr;26(2):137-41. doi: 10.1054/jhsb.2000.0487. PMID 11281665
- [Background] Upton AR, McComas AJ. The double crush in nerve entrapment syndromes. Lancet. 1973 Aug 18;2(7825):359-62. doi: 10.1016/s0140-6736(73)93196-6. No abstract available. PMID 4124532
- [Background] Leechavengvongs S, Malungpaishorpe K, Uerpairojkit C, Ng CY, Witoonchart K. Nerve Transfers to Restore Shoulder Function. Hand Clin. 2016 May;32(2):153-64. doi: 10.1016/j.hcl.2015.12.004. PMID 27094888
- [Background] Bhandari PS, Sadhotra LP, Bhargava P, Bath AS, Mukherjee MK, Bhatti T, Maurya S. Surgical outcomes following nerve transfers in upper brachial plexus injuries. Indian J Plast Surg. 2009 Jul;42(2):150-60. doi: 10.4103/0970-0358.59272. PMID 20368849
- [Background] Narakas AO, Hentz VR. Neurotization in brachial plexus injuries. Indication and results. Clin Orthop Relat Res. 1988 Dec;(237):43-56. PMID 3056647
- [Background] Waters PM, Smith GR, Jaramillo D. Glenohumeral deformity secondary to brachial plexus birth palsy. J Bone Joint Surg Am. 1998 May;80(5):668-77. doi: 10.2106/00004623-199805000-00007. PMID 9611027
- [Background] Buterbaugh KL, Shah AS. The natural history and management of brachial plexus birth palsy. Curr Rev Musculoskelet Med. 2016 Dec;9(4):418-426. doi: 10.1007/s12178-016-9374-3. PMID 27680748
- [Background] Terzis JK, Papakonstantinou KC. Management of obstetric brachial plexus palsy. Hand Clin. 1999 Nov;15(4):717-36. PMID 10563272
- [Background] Foad SL, Mehlman CT, Ying J. The epidemiology of neonatal brachial plexus palsy in the United States. J Bone Joint Surg Am. 2008 Jun;90(6):1258-64. doi: 10.2106/JBJS.G.00853. PMID 18519319
- See also: Related Info — https://clinicaltrials.gov